CLINICAL TRIAL: NCT04841720
Title: Phase I Clinical Study to Evaluate the Drug-drug Interaction Between HSK16149 Capsules and Metformin Hydrochloride Tablets in Healthy Subjects
Brief Title: A Study Evaluating Drug-Drug Interaction (DDI) Between HSK16149 Capsules and Metformin Hydrochloride Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK16149-103
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Diabetic Neuropathies; Diabetic Neuropathy Peripheral
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HSK16149 (Experimental): HSK16149（D1-D5）
  Interventions: Drug: HSK16149
- Metformin (Experimental): Metformin
  Interventions: Drug: Metformin Hydrochloride tablet
- HSK16149+Metformin (Experimental): HSK16149+Metformin
  Interventions: Drug: HSK16149+Metformin（phase 3）

INTERVENTIONS:
Drug: HSK16149 — HSK16149 capsules for single use: D1-D4 oral HSK16149 capsules 80 mg BID, D5 only oral HSK16149 capsules 80 mg in the morning on an empty stomach; wash-out period is about 4 days (D5-D8);
  Other Names: HSK16149（phase 1）
  Arms: HSK16149
Drug: Metformin Hydrochloride tablet — Metformin hydrochloride tablets for single use: D9-D11 oral metformin hydrochloride tablets 500 mg BID, D12 only take 500 mg metformin hydrochloride tablets in the morning on an empty stomach; wash-out period is about 4 days (D12-D15);
  Other Names: Metformin hydrochloride tablets（phase 2）
  Arms: Metformin
Drug: HSK16149+Metformin（phase 3） — Combined use of HSK16149 capsules and metformin hydrochloride tablets: D16-D19 oral metformin hydrochloride tablets 500 mg BID, D16-D19 oral HSK16149 80 mg BID; D20 oral metformin hydrochloride tablets 500 mg and HSK16149 capsules 80 mg in the morning on an empty stomach.
  Other Names: HSK16149 capsules and Metformin hydrochloride tablets
  Arms: HSK16149+Metformin

SUMMARY:
This study is a single-center, open, single-arm study, conducted in healthy Chinese populations, and plans to enroll 22 healthy adult subjects (the ratio of either sex is not less than 1/3).

DETAILED DESCRIPTION:
All subjects received the following drugs:

Phase 1-HSK16149 capsules for single use: D1-D4 oral HSK16149 capsules 80 mg BID, D5 only oral HSK16149 capsules 80 mg in the morning on an empty stomach; wash-out period is about 4 days (D5-D8); Phase 2-Metformin hydrochloride tablets for single use: D9-D11 oral metformin hydrochloride tablets 500 mg BID, D12 only take 500 mg metformin hydrochloride tablets in the morning on an empty stomach; wash-out period is about 4 days (D12-D15); Phase 3-Combined use of HSK16149 capsules and metformin hydrochloride tablets: D16-D19 oral metformin hydrochloride tablets 500 mg BID, D16-D19 oral HSK16149 80 mg BID; D20 oral metformin hydrochloride tablets 500 mg and HSK16149 capsules 80 mg in the morning on an empty stomach.

ELIGIBILITY:
Inclusion Criteria:

1. 18-50 years old (including 18 and 50 years old), healthy male or female;
2. Weight: male ≥50 kg, female ≥45kg; body mass index (BMI) in the range of 19-28kg/m2 (including 19 and 28);
3. Serum creatinine during the screening period is within the normal range, or creatinine clearance rate (CCr) ≥80mL/min;
4. Physical examination, vital signs, 12-lead electrocardiogram (ECG), chest X-ray (posterior anterior position), and laboratory examination indicators are normal or abnormal and have no clinical significance;
5. Agree to have no birth plan and be able to take reliable contraceptive measures within 3 months after the end of the trial; Be able to communicate well with researchers, fully understand the purpose and requirements of this trial, voluntarily participate in clinical trials and sign written informed consent.

Exclusion Criteria:

1. Those who are known to have a history of allergies, allergic diseases or allergies to the research preparation and any of its ingredients or related preparations, or those who have a history of pregabalin or gabapentin allergy;
2. Those who have special requirements for diet and cannot comply with a unified diet;
3. Those who have had angioedema in the past;
4. Clinically significant dizziness or vertigo, or a history of inner ear diseases known to cause dizziness or vertigo;
5. QTcF>450 milliseconds (msec) found in the screening period inspection;
6. People with insomnia, anxiety disorder, depression disorder or other mental disorders;
7. Those who use any caffeine-rich food or drink (coffee, tea, cola, chocolate, etc.) within 48 hours before the first administration of the test drug, or who do not agree to prohibit the use of any caffeine-rich food or drink during the test period ；
8. Any disease history or current disease that may affect the safety evaluation of subjects or the internal process of experimental drugs, including the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, immunology, Psychiatry, metabolic abnormalities, gastrointestinal surgery (except appendicitis surgery), etc.;
9. Those who donate blood or lose blood ≥400 mL or have blood transfusion within 3 months before the first administration of the test drug;
10. Any drug that inhibits or induces liver drug-metabolizing enzymes (such as inducers barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole) has been used within 30 days before the first administration of the test drug; Serotonin reuptake inhibitor (SSRI) antidepressants, cimetidine, diltiazem macrolides, nitroimidazoles, sedative hypnotics, verapamil, fluoroquinolones, antihistamines), or Any prescription drugs, over-the-counter drugs and herbal medicines other than the above-mentioned drugs were taken within 14 days prior to the administration of the test drugs;
11. Those who have participated in other drug clinical trials within 3 months before the first administration of the experimental drug;
12. At this stage or have been drug users, or those who have been screened positive for drug abuse (screening items include: morphine, tetrahydrocannabinolic acid, methamphetamine, dimethylenedioxyamphetamine, Ketamine and cocaine);
13. Alcoholics or frequent alcoholics in the 3 months before the test, that is, drinking more than 21 units of alcohol per week (1 unit = 360mL beer or 45 mL 40% alcoholic spirits or 150 mL wine), or alcohol exhalation Test value> 0mg/ml;
14. Smokers or those who smoked more than 10 cigarettes per day within 3 months before the first administration, or who could not comply with the ban on smoking during the trial period;
15. One or more of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, syphilis antibody or human immunodeficiency virus (HIV) antibody is positive;
16. Women during pregnancy or lactation;Researchers believe that subjects have poor compliance or other factors that are not suitable for participating in this trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Cmax | -30 minutes before administration until 24 hours after administration
  Peak concentration
AUC0-t, AUC0-∞ | -30 minutes before administration until 24 hours after administration
  Area under the concentration-time curve
Tmax | -30 minutes before administration until 24 hours after administration
  time to peak observed

SECONDARY OUTCOMES:
AE/serious AE | From screening up to 6 weeks
  Adverse event/serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Mingxia Wang, PhD, Study Director — Medical Ethics Committee of theThe fourth hospital of Hebei Medical University
Locations (1):
- The fourth hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No